CLINICAL TRIAL: NCT00003431
Title: Pilot Study of FLT3 Ligand Prior to Resection of Hepatic Metastases of Colorectal Cancer
Brief Title: Flt3L in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066457; DUMC-98032; NCI-G98-1454
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; lung metastases; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms | interventions — flt3 ligand protein

INTERVENTIONS:
Biological: recombinant flt3 ligand

SUMMARY:
RATIONALE: Flt3L may stimulate a person's immune system and help kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of flt3L given to patients before undergoing surgery to remove metastases from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the safety and feasibility of administering flt3 ligand to patients with hepatic metastases from colorectal cancer prior to surgical resection.

OUTLINE: Patients receive flt3 ligand subcutaneously for 14 days followed by 14 days of rest. This course of therapy may be repeated for a total of 3 courses. Leukapheresis is performed on day 15 of the last course of Flt3 ligand. Patients undergo restaging and metastasis resection. Patients are followed every 3 months for the first year, every 6 months for the second year, and yearly thereafter.

PROJECTED ACCRUAL: This study will accrue 12 patients in 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic colon cancer expressing carcinoembryonic antigen (CEA) At least 50% of tumor cells must express CEA with at least moderate intensity Resectable hepatic metastases or other site of metastatic colon cancer that is resectable (e.g., lung metastases)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 6 months Hematopoietic: Absolute neutrophil count at least 1000/mm3 Absolute lymphocyte count at least 1000/mm3 Hemoglobin at least 9 mg/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL No hepatic disease Renal: Creatinine less than 2.5 mg/dL Cardiovascular: No ongoing cardiac disease No New York Heart Association class III or IV heart disease Pulmonary: No ongoing pulmonary disease such as: Asthma Chronic obstructive pulmonary disease (COPD) Active radiation- or drug-induced pneumonitis Other: Not pregnant or nursing Fertile patients must use effective contraception No history of autoimmune disease such as but not limited to: Inflammatory bowel disease Systemic lupus erythematosus Ankylosing spondylitis Scleroderma Type I diabetes Multiple sclerosis No other serious ongoing chronic or acute illness No medical or psychological impediment to study compliance No concurrent or prior second malignancy except: Nonmelanoma skin cancer Controlled superficial bladder cancer within the last 5 years No active or chronic infection including: Urinary tract infection HIV Viral hepatitis

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No concurrent chemotherapy Endocrine therapy: No concurrent corticosteroids No concurrent hormone therapy Radiotherapy: No concurrent radiation therapy Surgery: No specified Other: No immunosuppressives such as: Azathioprine Cyclosporine A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Morse, MD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States